CLINICAL TRIAL: NCT06217263
Title: Effect of Vibration and Cold Application on Chest Tube Removal Pain After Coronary Artery Bypass Graft Surgery
Brief Title: Effect of Vibration and Cold Application on Chest Tube Removal Pain After CABG
Acronym: CABG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Oyku Kara, Surgical Nursing Research Assistant (Master), Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3435-123
Record Dates: First submitted 2023-12-24; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Pain, Procedural; Pain, Postoperative; Coronary Artery Bypass Surgery; Chest Tubes
Keywords: Pain; Postoperative pain; Coronary artery bypass surgery; Chest tube pain; vibration; cold application; pain management; nursing
MeSH Terms: conditions — Pain, Procedural; Pain, Postoperative; Pain; Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vibration (Experimental): After coronary artery bypass graft surgery, patients will receive routine monitoring, pharmacological treatment and nursing care in the unit where the research is conducted. The vibration device will be placed in the upper quadrant proximal to the patient's drain tube entrance. Care will be taken to ensure that the point where the vibration device is placed is the same as the vibration device placement point in the vibration and cold application group. 10 minutes after the application, the patient's skin temperature will be measured and the vibration device will be pulled above the chest tube insertion area.
  Interventions: Device: Vibration device
- Vibration & Cold application (Experimental): After coronary artery bypass graft surgery, patients will receive routine monitoring, pharmacological treatment and nursing care in the unit where the research is conducted. Cold gel pack will be placed around the patient's chest tube insertion area. In order to optimize the effect of cold, the cold application will not exceed 20 minutes and the temperature of the skin will not fall below 12 ℃. At the 10th minute of cold application, the vibration device will be placed proximal to the chest tube, over the upper area of the cold gel pack. At the 20th minute of the application, the patient's skin temperature will be measured and the cold applied vibration device will be pulled above the chest tube insertion area.
  Interventions: Other: Vibration device&Cold application pack
- Control (No Intervention): After coronary artery bypass graft surgery, patients will receive routine monitoring, pharmacological treatment and nursing care in the unit where the research is conducted. In the control group, the processes and monitoring in the application groups will be continued in the same period without the application.

INTERVENTIONS:
Device: Vibration device — Vibracool vibration device from Pain Care Labs will be used.
  Arms: Vibration
Other: Vibration device&Cold application pack — Pain Care Labs' Vibracool vibration device and cold gel pack will be used.
  Arms: Vibration & Cold application

SUMMARY:
After cardiothoracic surgery, a chest tube is placed in patients to maintain hemodynamic stability and cardiopulmonary function by evacuating air, blood, and fluid accumulated in the pleural, pericardial, or mediastinal space, and to prevent undesirable conditions such as pneumothorax, hemothorax, and pleural effusion. Chest tube removal (CTR); it is an experience that can cause moderate or severe pain and anxiety in patients due to friction and separation from the endothelium and other surrounding tissues in the entry area of the tube. Analgesic methods are often preferred in pain management. However, research reveals that patients experience pain during CTR despite the use of analgesics and anesthetics. Although pharmacological agents are the most commonly used method for pain relief during CTR, studies report that the response to pharmacological treatment is variable and may be inadequate for pain management during and after CTR, making pain management difficult. Considering that procedure-related anxiety disrupts the physiological and emotional state of the patient and the side effects and possible complications of analgesics used in pain management, such as respiratory distress and nausea, the importance of nurses' use of non-drug methods in reducing pain during CTR increases This research was designed as a randomized controlled experimental study to determine the effect of vibration and cold application on pain and anxiety associated with chest tube removal after coronary artery bypass graft surgery. The research was planned to be conducted in the Cardiovascular Surgery Intensive Care Unit and Surgical Services of a Thoracic and Cardiovascular Surgery Training and Research Hospital in Istanbul between January 2024 and January 2025. Patients' pain will be evaluated using VAS, blood pressure, and respiratory rate using a patient monitor, pulse and oxygen saturation using a pulse oximeter device, and the temperature of cold application gels using a digital infrared thermometer. All data will be collected by the same researcher, with the same tools and methods. A "data form" developed in line with the literature and STAI I-II (State and Trait Anxiety Scale) will be used as data collection tools.

DETAILED DESCRIPTION:
In patients undergoing Coronary Artery Bypass Graft (CABG) surgery, opening a sternotomy, cutting the intercostal nerves along the incision line, turning in bed, breathing, deep breathing, coughing, pleural irritation associated with the chest tube and removal of the chest tube are situations that cause pain. 74% of patients experience moderate to severe pain despite pharmacological treatment. After cardiothoracic surgery, a chest tube is placed in patients to maintain hemodynamic stability and cardiopulmonary function by evacuating air, blood, and fluid accumulated in the pleural, pericardial, or mediastinal space, and to prevent undesirable conditions such as pneumothorax, hemothorax, and pleural effusion. Chest tube removal (CTR); it is an experience that can cause moderate or severe pain and anxiety in patients due to friction and separation from the endothelium and other surrounding tissues in the entry area of the tube. Analgesic methods are often preferred in pain management.However, research reveals that patients experience pain during CTR despite the use of analgesics and anesthetics. Although pharmacological agents are the most commonly used method for pain relief during CTR, studies report that the response to pharmacological treatment is variable and may be inadequate for pain management during and after CTR, making pain management difficult. Considering that procedure-related anxiety disrupts the physiological and emotional state of the patient and the side effects and possible complications of analgesics used in pain management, such as respiratory distress and nausea, the importance of nurses' use of non-drug methods in reducing pain during CTR increases. In this context, the use of cold and vibration applications, which do not require invasive intervention, involves minimal risk, and can be easily applied by nurses, are practices that can contribute to the improvement of patient outcomes by reducing the pain experienced by the patient during CTR.

In the study, in order to determine the effect of vibration and cold application on pain and anxiety associated with chest tube removal after coronary artery bypass graft surgery, the calculation (d-value) method developed by Cohen was used to calculate the effect size to be used to determine the sample size to be included in the study. To determine the d value, which is the effect size index, the findings of the study reported by Yurdanur and Khorshid in 2010, which investigated the effect of cold application combined with standard analgesics on pain and anxiety during chest tube removal in patients undergoing thoracic surgery, were used. The effect size to be used in the research was calculated as d = 0.329. In this context, for the quantitative difference test (ANOVA test) between the three groups, d = 0.329, 95% confidence level (1-α), 80% test power (1-β) and 31 samples in each group using the G-power (version 3.1) package program. It was envisaged that a total of 93 participants would be taken as the sample group. A simple computer-assisted randomization method was used to distribute the groups homogeneously. For this purpose, the functions available on the website "https://www.random.org/integer-sets" were used.

Ethical permission was received for the research from the Clinical Research Ethics Committee (Decision No: 239, Date: 04.07.2023). Device usage permission is awaited from the Turkish Medicines and Medical Devices Agency.

ELIGIBILITY:
Inclusion Criteria:

* A chest tube was placed for the first time
* ASA (American Society of Anesthesiology) classification I and II
* Those between the ages of 40-65
* Conscious, oriented and cooperative
* Patients who agree to participate in the research verbally and in writing after being informed about the research

Exclusion Criteria:

* Having a chest tube for more than 72 hours
* More than one chest tube entry and removed at the same time
* A chest tube was removed from the area close to the sternotomy line
* Having compromised skin integrity (burn, laceration, scar, inflammation, infection, erythema) around the chest tube and in the application area
* Having a history of thoracotomy
* Those who are intubated
* Those with cold urticaria
* Under the influence of anesthesia or analgesia
* Complications developed during or after surgical intervention
* Those who do not speak Turkish and have hearing and vision problems
* Having a diagnosed psychiatric disease or mental problem
* Having a body mass index ≥30
* Patients who participated in another clinical trial during the same period

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain using the Visual Analog Scale | Change from baseline (before application) and 15-minute change after application
  Pain associated with chest tube removal. Visual Analog Scale (VAS) is the most frequently used and simplest to use scale. In the scale with numbers between 0-10, "0" defines painlessness and "10" defines the most severe pain.
  In order to define the numerical value of the patient's pain/anxiety severity, the patient is asked to mark the ruler consisting of a 10 cm line, and the patient's pain severity score is determined as a result of the measurement.
  The scale consists of five parts. Each of the sections is in the range of 2 points. '0' points - no pain, '1-2 points, very mild pain', '3-4 points, mild pain', '5-6 points, moderate pain', '7-8 points, severe pain' means '9-10 points, excruciating pain'.
Assessment of pain using the The State-Trait Anxiety Inventory Scale | Change from baseline (before application) and 15-minute change after application
  State-Trait Anxiety Inventory (STAI); STAI-I was developed by Spielberger in 1970. The scale consists of 20 items. The answers range from 1-4. The total point value obtained from the scale is between 20-80. A high score indicates a high level of anxiety. STAI 2 Trait Anxiety Scale; It aims to measure how the individual feels, that is, his trait anxiety, regardless of the situation and conditions he is in. In answering the state anxiety scale; choosing one of the options "Not at all", "A little", "A lot", "Totally" according to the level of severity of the feelings, behaviors or thoughts expressed by the items; In answering the trait anxiety scale, it is required to select and mark one of the options "Almost Never", "Sometimes", "Very Often" and "Almost Always" according to the frequency level of the feelings, behaviors or thoughts expressed by the items.obtaining informed consent. The state anxiety level will be evaluated before and after the interventions.

SECONDARY OUTCOMES:
Pulse rate | Change from baseline (before application) and 15-minute change after application
  The pulse rate will be evaluated with the clinical patient monitor.
Oxygen saturation | Change from baseline (before application) and 15-minute change after application
  The oxygen saturation will be evaluated with the clinical patient monitor.
Systolic and diastolic blood pressure | Change from baseline (before application) and 15-minute change after application
  Systolic and diastolic blood pressure will be assessed with a cuffed clinical patient monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Oyku Kara, MSc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- IstanbulUC, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No